CLINICAL TRIAL: NCT04134806
Title: Evaluation of a Navigation Experiment in the Gait Real-Time Analysis Interactive Lab: Gait Analysis by Induced Disorientation in a VR Environment
Brief Title: Gait Analysis by Induced Disorientation in a VR Environment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Rostock (Other)
Collaborators: University of Rostock (Other); German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Stefan Teipel, Prof. Dr., University Medical Center Rostock
Organization: University of Rostock (Other)
Other Study IDs: A 2019-0062
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Disorientation; Young Adults; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Confusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7.5 millilitre blood sample for Apolipoprotein E4 (ApoE4) analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young Adults: Neurologically healthy young adults between ages 18 and 40
- Older Adults: Neurologically healthy older adults between ages 60 and 85
- Mild Cognitive Impairment/Mild Dementia: Older adults between ages 60 and 85 with Mild Cognitive Impairment or Mild Dementia

SUMMARY:
The aim of the study is to investigate whether the effect of disorientation on physical motion and gait among dementia patients, can be reliably measured in a laboratory environment, by means of a virtual reality (VR) experimental setup.

DETAILED DESCRIPTION:
Challenges in wayfinding and orientation are early symptoms of MCI and dementia. These deficits decrease mobility which again leads to further cognitive decline. In a field study, we developed a pattern recognition model of disorientated behaviour based on accelerometric data. However, it is questionable if phases of disorientation also affect gait parameters. Furthermore, there is growing evidence that impaired cognitive functioning is associated with changes in gait performance, e.g. gait variability, measured in dual-task walking conditions. Increases in heart rate and skin conductance have also been reported during instances of disorientation.

Hence, We implemented a 3D environment of a familiar city centre in the GRAIL, which combines a fully instrumented treadmill with a synchronized VR environment. We record gait parameters through the motion capture system, and accelerometric and physiological data using wearable sensors (movisens), for comparability with the SiNDeM field study. Young and old healthy adults will participate in the first phase of the study, while Mild dementia or MCI patients will participate in the later phases. Phases of disorientation will be induced by changing the virtual environment.We aim to assess gait, accelerometric and physiological parameters during instances of disorientation, using the GRAIL (Gait Real-Time Analysis Interactive Lab, Motekforce Link).

The results will further enable the automatic detection of disorientation based on gait parameters, physiological and accelerometric data. This is necessary for the development of a situation-aware assistive system which supports persons with dementia in autonomous outdoor mobility.

ELIGIBILITY:
Inclusion Criteria:

* Within the required age bracket
* Mobile
* Dementia

Exclusion Criteria:

* Other neurological conditions besides dementia
* Inability to understand task instructions, deaf-mute, blindness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young adults, healthy older adults and older adults with mild cognitive impairment or mild dementia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Spatial disorientation | Up to 3 years from start of the study
  Incidences of disorientation will be captured in a video record during the experiment, and then later identified in an off-line annotation procedure using a customized annotation scheme

SECONDARY OUTCOMES:
Gait variability | Up to 3 years from start of the study
  Incidences of change in gait pattern will be measured using the gait capturing system of the GRAIL (gait real-time analysis interactive lab)
Spatial orientation ability | Up to 3 years from start of the study
  Older adult participants' spatial orientation ability will be evaluated using the Perspective taking spatial orientation test (PTSOT). No predefined range. Lower scores indicate better spatial orientation ability. Formula: sum of true angles - sum of expressed angles
Heart rate variability | Up to 3 years from start of the study
  Rate of change in heart rate will be measured using a wearable electrocardiographic sensor
Skin conductance | Up to 3 years from start of the study
  Rate of change in electrodermal response will be measured using a wearable electrodermal activity sensor
Accelerometery | Up to 3 years from start of the study
  Incidences of change in walking pattern will be measured using accelerometers
Apolipoprotein E4 status | Up to 3 years from start of the study
  Presence of the variants Apo-E2, E3 and -E4 in the blood samples
Visuospatial function | Up to 3 years from start of the study
  Older adult participants' visual constructive ability will be evaluated using the figure copy part of the Rey-Osterrieth complex figure test (ROCF). Higher scores indicate better visual constructive ability. Range 0-31
Memory function | Up to 3 years from start of the study
  Older adult participants' spatial memory will be evaluated using the figure recall part of the Rey-Osterrieth complex figure test (ROCF). Higher scores indicate better memory. Range 0-31
Executive function | Up to 3 years from start of the study
  Older adult participants' executive function will be evaluated using the Trail making test (TMT A/B). Lower scores indicate better executive function. No predefined range

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J. Teipel, Prof. Dr., Principal Investigator — University Medical Center Rostock
Locations (1):
- Clinic and Polyclinic for Psychosomatics and Psychotherapeutic Medicine, University Medical Center Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaat S, Koldrack P, Yordanova K, Kirste T, Teipel S. Real-Time Detection of Spatial Disorientation in Persons with Mild Cognitive Impairment and Dementia. Gerontology. 2020;66(1):85-94. doi: 10.1159/000500971. Epub 2019 Jul 30. PMID 31362286
- [Background] Yordanova K, Koldrack P, Heine C, Henkel R, Martin M, Teipel S, Kirste T. Situation Model for Situation-Aware Assistance of Dementia Patients in Outdoor Mobility. J Alzheimers Dis. 2017;60(4):1461-1476. doi: 10.3233/JAD-170105. PMID 29060937
- [Derived] Amaefule CO, Ludtke S, Kirste T, Teipel SJ. Effect of Spatial Disorientation in a Virtual Environment on Gait and Vital Features in Patients with Dementia: Pilot Single-Blind Randomized Control Trial. JMIR Serious Games. 2020 Oct 8;8(4):e18455. doi: 10.2196/18455. PMID 33030436